CLINICAL TRIAL: NCT07072689
Title: A Single-centre Study Evaluating the Performance and Acceptance of the Hilo Band Cuffless Blood Pressure Medical Device in the Normo-, Hypo- and Hyper-tensive Young Population: a Comparison With the 24-h Ambulatory Blood Pressure Monitoring (ABPM)
Acronym: IPSI-HYPE-001
Status: Not yet recruiting | Type: Observational
Sponsor: Simonetti Giacomo (Other)
Responsible Party: Sponsor-Investigator, Simonetti Giacomo, Prof. Dr. med, Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Other Study IDs: IPSI-HYPE-001
Record Dates: First submitted 2025-06-11; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Hypertension
Keywords: Aktiia; 24-h ABPM; hypertension; young; blood pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Population 2: No indications for blood pressure measurements
- Population 1: Indications to receive blood pressure measurement of 24-hours

SUMMARY:
Hypertension is one of the main risk factors for the onset of cardiovascular diseases. It is often silent, and most individuals are unaware they have it.

The 24-hour Ambulatory Blood Pressure Monitoring (24-hour ABPM) device allows for continuous blood pressure monitoring over a 24-hour period and is currently considered the gold standard for diagnosing hypertension. However, it is expensive, time-consuming for healthcare personnel, bulky, and often uncomfortable to wear-especially during the night.

Recently, other blood pressure monitoring devices have entered the market. One of them is the Aktiia bracelet, renamed as Hilo band as of 8 april 2025, (Hilo band SA, Neuchâtel, Switzerland), CE-marked, which estimates blood pressure and heart rate using a pulse wave analysis (PWA) technique. Hilo band is non-invasive, comfortable to wear, and allows for long-term blood pressure monitoring.

However, there is insufficient data to support the use of Hilo band in healthcare settings for the diagnosis and monitoring of hypertension. In one study, Hilo band was compared to the 24-hour ABPM only for daytime blood pressure readings in a population enrolled in a cardiac rehabilitation program, and thus was not tested in apparently 'healthy' individuals who may be hypertensive. Another study assessed Hilo band's performance compared to double auscultation in older adults aged 65 to 85 years in different body positions (sitting, standing, and lying down), and therefore did not include a younger population.

In our research project, we aim to evaluate the performance of Hilo band compared to 24-hour ABPM in a younger population, considering both daytime and nighttime blood pressure measurements.

DETAILED DESCRIPTION:
This research project is a single-center non-interventional performance study of San Giovanni Hospital in Bellinzona comparing the systolic and diastolic blood pressure measurement of Hilo band with the systolic and diastolic blood pressure measurement of the 24-h ABPM of 40 young participants between 21 and 35 years of age.

ELIGIBILITY:
Inclusion Criteria:

Population 2:

* Informed Consent signed by the subject
* 21-35 years of age
* Functional internet phone connection
* Negative pregnancy test, ongoing anti-conceptive treatment or declaration of the subject not being pregnant

Population 1:

* Informed Consent signed by the subject
* 21-35 years of age
* Clinical indication for receiving a 24-hour blood pressure measurement
* Functional internet phone connection
* Negative pregnancy test, ongoing anti-conceptive treatment or declaration of the subject not being pregnant

Exclusion Criteria for both population 1 and 2:

* Allergies to silicone
* Atrial fibrillation
* Subjects with arrhythmia
* Patients suffering from pathologies that systematically reduce peripheral perfusion including Raynaud's disease, diabetes, renal dysfunctions (eGFR < 30mL / min / 1.73 m2), untreated hyper-/ hypothyroidism, pheochromocytoma, or arteriovenous fistula
* Interarm Systolic Blood Pressure (SBP) difference over 10% or Diastolic Blood Pressure (DBP) difference over 10%
* Arm paralysis
* Amputated upper limb
* Arm trembling or shivering
* Upper arm circumference > 64 cm
* Wrist circumference > 22 cm
* Exfoliative skin diseases and lymphoedema or damaged/injured skin at the wrist
* Pregnant women
* Individuals with lack of judgment/mental illness
* Sleepwalking and severe insomnia
* Pica disorder

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This is a single-centre non-interventional performance research project investigating the performance of Hilo band in two different study populations: population 1 and population 2.
  In population 1, we will recruit young participants between 21 and 35 years of age that come to our San Giovanni Hospital in Bellinzona with indication to receive a 24-hour BPM.
  On the other hand, in population 2, we will recruit healthy, voluntary individuals between 21 and 35 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the 24-hour performance of Hilo band in measuring diastolic and systolic blood pressure values in young subjects of 21-35 years of age. We will use the 24h ABPM as a reference method | 24 hours
  To assess our primary endpoint, the 24-hour systolic and diastolic pressure averages (including waking and sleeping hours) of Hilo band will be compared to the 24-hour systolic and diastolic pressure averages of the 24-h ABPM, respectively. A similar performance of the two devices is defined as a standard deviation from the 24-hour (including waking and/or sleeping hours) average systolic and/or diastolic pressure values of maximum 10 mmHg, as reported in previous studies.
  We will consider valid and include in the analysis 24-h ABPM recordings lasting ≥22 hours with ≥80% of successful readings, and cumulative recording gaps no greater than 2 hours.
  On the other hand, Hilo band's blood pressure recordings are considered valid if at least 24 measurements are recorded during the 24 hours period.

SECONDARY OUTCOMES:
Assessing the consistency of the performance of Hilo band in measuring systolic and diastolic blood pressure values in young subject of 21-35 years of age over a 3-day period with the 24-h ABPM as a reference method | 3 days
  The 72-hour systolic and diastolic pressure averages (including waking and sleeping hours) of Hilo band will be compared to the 24-hour systolic and diastolic pressure averages of the 24-h ABPM, respectively. A similar performance of the two devices is defined as a difference in the average 72-hour (for Hilo band) and 24-hours (for the 24-h ABPM) systolic and diastolic pressure values (including waking and sleeping hours) of up to 10 mmHg, as reported in previous studies.
  We will consider valid and include in the analysis 24-h ABPM recordings lasting ≥22 hours with ≥80% of successful readings, and cumulative recording gaps no greater than 2 hours.
  On the other hand, Hilo band blood pressure recordings are considered valid if at least 24 measurements are recorded per day/24-hours, for a total of at least 72 measurements recorded during the 3 days/72 hours period.
Evaluate the performance of Hilo band in effectively classifying hypertension in young subjects of 21-35 years of age with the 24-h ABPM as a reference method. | 3 days
  We assess Hilo band's performance in classifying hypertensive and normotensive subjects as effective if Hilo band correctly classifies 90% of hypertensive subjects and 90% normotensive subjects, respectively. We define hypertensive and normotensive individuals as follows:
  Hypertension for systolic and diastolic blood pressure measurement of Hilo band and 24-h ABPM:
  * 24-h average: ≥ 130 mmHg and/or ≥80 mmHg
  * Day time (or awake) average: ≥ 135 mmHg and/or ≥ 85 mmHg
  * Night time (or sleep) average: ≥ 120 mmHg and/or ≥ 70 mmHg
  Normotension for systolic and diastolic blood pressure measurement of Hilo band and 24-h ABPM:
  * 24-h average: < 130 mmHg and/or < 80 mmHg
  * Day time (or awake) average: < 135 mmHg and/or < 85 mmHg
  * Night time (or sleep) average: < 120 mmHg and/or < 70 mmHg
Evaluate the degree of satisfaction of the use of the Hilo band by study participants and physicians with the 24-h ABPM as a reference method. | 3 days
  The questionnaires we use to assess the degree of satisfaction with the use of Hilo band by the physicians and participants consist of two types of questions: questions with yes/no answers and questions with answers ranging from 1 (lowest satisfaction) to 5 (highest satisfaction). We define the degree of satisfaction with the use of Hilo band by the participants and physicians as follows:
  * For questions with yes/no answers:
    1. 0-49% of total yes answers: participants and physicians not satisfied
    2. 50-69% of total yes answers: participants and physicians fairly satisfied
    3. 70-100% of total yes answers: participants and physicians very satisfied
  * For questions with answers from 1 to 10:
    1. Average of answers < 2.75: participants and physicians not satisfied
    2. Average of answers between 2.75 and 3.75: participants and physicians fairly satisfied
    3. Average of answers > 3.75: participants and physicians very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Simonetti, Prof. Dr. med, Principal Investigator — Ente Ospedaliero cantonale (EOC)
Locations (1):
- Ente Ospedaliero Cantonale, Bellinzona, Switzerland